CLINICAL TRIAL: NCT00005536
Title: Genetic Analysis of Human Hypertensive End Stage Renal Disease (H-ESRD)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5069; R01HL056266 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2005-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Kidney Failure, Chronic
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Kidney Failure, Chronic

SUMMARY:
To identify genes causing hypertensive end-stage renal disease (H-ESRD) in high risk African-American populations

DETAILED DESCRIPTION:
BACKGROUND:

Although hypertension is a predisposing factor for end stage renal disease, the underlying hypothesis of this study was that in select African-American families genetic factors predisposed them to develop ESRD in the face of hypertension. An inherited basis for H-ESRD was supported by familial clustering of H-ESRD among African Americans that could not be explained by socioeconomic status, access to medical care, and the prevalence of diabetes and hypertension.

DESIGN NARRATIVE:

DNA samples were collected, identified, and clinically characterized from African-American sib-pairs (and other family members with hypertensive end-stage renal disease). This aspect of the study was based on the fact that Dr. Freedman, the principal investigator, had already developed a unique "family history of end-stage renal disease" database independently funded by the End-Stage Renal Disease Network Six. This registry served as a very large and unique collection of African-American end-stage renal disease patients. He began with a candidate gene approach for linkage to hypertensive end-stage renal disease in his patient samples using a variety of growth factor genes, genes involved in sodium transport and vascular tone, as well as human homologues of rodent genes that had, or were to be identified in the future as contributing to ESRD in that organism. If this initial first pass of candidate genes failed to demonstrate linkage to hypertensive end-stage renal disease, a systematic genome-wide scan was to be performed with available simple sequence length polymorphisms (SSLP) and other polymorphic markers. Hypertensive end-stage renal disease is a condition of enormous clinical and economic importance and identification of associated or causative renal-failure genes would form a genetic basis for the detection of high-risk individuals and assist in development of intervention and treatment strategies to prevent this condition.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-07; Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry Freedman — Wake Forest University

REFERENCES:
- [Background] Price JA, Fossey SC, Sale MM, Brewer CS, Freedman BI, Wuerth JP, Bowden DW. Analysis of the HNF4 alpha gene in Caucasian type II diabetic nephropathic patients. Diabetologia. 2000 Mar;43(3):364-72. doi: 10.1007/s001250050055. PMID 10768098
- [Background] Freedman BI, Soucie JM, Chapman A, Krisher J, McClellan WM. Racial variation in autosomal dominant polycystic kidney disease. Am J Kidney Dis. 2000 Jan;35(1):35-9. doi: 10.1016/S0272-6386(00)70298-8. PMID 10620541
- [Background] Yu H, Freedman BI, Rich SS, Bowden DW. Human Na+/H+ exchanger genes : identification of polymorphisms by radiation hybrid mapping and analysis of linkage in end-stage renal disease. Hypertension. 2000 Jan;35(1 Pt 1):135-43. doi: 10.1161/01.hyp.35.1.135. PMID 10642288
- [Background] Freedman BI, Soucie JM, Stone SM, Pegram S. Familial clustering of end-stage renal disease in blacks with HIV-associated nephropathy. Am J Kidney Dis. 1999 Aug;34(2):254-8. doi: 10.1016/s0272-6386(99)70352-5. PMID 10430971
- [Background] Yu H, Sale M, Rich SS, Spray BJ, Roh BH, Bowden DW, Freedman BI. Evaluation of markers on human chromosome 10, including the homologue of the rodent Rf-1 gene, for linkage to ESRD in black patients. Am J Kidney Dis. 1999 Feb;33(2):294-300. doi: 10.1016/s0272-6386(99)70303-3. PMID 10023641
- [Background] Yu H, Bowden DW, Spray BJ, Rich SS, Freedman BI. Identification of human plasma kallikrein gene polymorphisms and evaluation of their role in end-stage renal disease. Hypertension. 1998 Apr;31(4):906-11. doi: 10.1161/01.hyp.31.4.906. PMID 9535413
- [Background] Ramerstorfer J, Furtmuller R, Vogel E, Huck S, Sieghart W. The point mutation gamma 2F77I changes the potency and efficacy of benzodiazepine site ligands in different GABAA receptor subtypes. Eur J Pharmacol. 2010 Jun 25;636(1-3):18-27. doi: 10.1016/j.ejphar.2010.03.015. Epub 2010 Mar 19. PMID 20303942
- [Background] Freedman BI, Yu H, Anderson PJ, Roh BH, Rich SS, Bowden DW. Genetic analysis of nitric oxide and endothelin in end-stage renal disease. Nephrol Dial Transplant. 2000 Nov;15(11):1794-800. doi: 10.1093/ndt/15.11.1794. PMID 11071967
- [Background] Yu H, Anderson PJ, Freedman BI, Rich SS, Bowden DW. Genomic structure of the human plasma prekallikrein gene, identification of allelic variants, and analysis in end-stage renal disease. Genomics. 2000 Oct 15;69(2):225-34. doi: 10.1006/geno.2000.6330. PMID 11031105
- [Background] Fossey SC, Mychaleckyj JC, Pendleton JK, Snyder JR, Bensen JT, Hirakawa S, Rich SS, Freedman BI, Bowden DW. A high-resolution 6.0-megabase transcript map of the type 2 diabetes susceptibility region on human chromosome 20. Genomics. 2001 Aug;76(1-3):45-57. doi: 10.1006/geno.2001.6584. PMID 11549316
- [Background] Freedman BI, Soucie JM, Kenderes B, Krisher J, Garrett LE, Caruana RJ, McClellan WM. Family history of end-stage renal disease does not predict dialytic survival. Am J Kidney Dis. 2001 Sep;38(3):547-52. doi: 10.1053/ajkd.2001.26851. PMID 11532687
- [Background] Gitter J, Langefeld CD, Rich SS, Pedley CF, Bowden DW, Freedman BI. Prevalence of nephropathy in black patients with type 2 diabetes mellitus. Am J Nephrol. 2002 Jan-Feb;22(1):35-41. doi: 10.1159/000046672. PMID 11919401
- [Background] Fan ZJ, Lackland DT, Kenderes B, Krisher J, Freedman BI. Impact of birth weight on familial aggregation of end-stage renal disease. Am J Nephrol. 2003 Mar-Apr;23(2):117-20. doi: 10.1159/000068037. PMID 12481151
- [Background] Freedman BI, Rich SS, Yu H, Roh BH, Bowden DW. Linkage heterogeneity of end-stage renal disease on human chromosome 10. Kidney Int. 2002 Sep;62(3):770-4. doi: 10.1046/j.1523-1755.2002.00534.x. PMID 12164858
- [Background] Yu H, Song Q, Freedman BI, Chao J, Chao L, Rich SS, Bowden DW. Association of the tissue kallikrein gene promoter with ESRD and hypertension. Kidney Int. 2002 Mar;61(3):1030-9. doi: 10.1046/j.1523-1755.2002.00198.x. PMID 11849458
- [Background] Satko SG, Langefeld CD, Daeihagh P, Bowden DW, Rich SS, Freedman BI. Nephropathy in siblings of African Americans with overt type 2 diabetic nephropathy. Am J Kidney Dis. 2002 Sep;40(3):489-94. doi: 10.1053/ajkd.2002.34888. PMID 12200799